CLINICAL TRIAL: NCT04880915
Title: Investigation of The Effect Of Fıve Different Methods On Surgical Smoke Protection Experimental Research
Brief Title: Effect of Fıve Different Methods On Smoke
Acronym: SurgicalSmok
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Burcak Sahin Koze, Principal Investigator, Ege University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Experimental
Record Dates: First submitted 2021-04-24; First posted 2021-05-11 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Exposure Occupational
Keywords: Surgical smoke; operating room; employee safety; nursing
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMOKE PROTECTION (Experimental): Pre- and post-operative blood and urine samples of the surgical team (surgeon, surgical resident, anaesthesiologist, scrub nurse, circulating nurse, support staff and researcher), who worked in the standard practice, and the use of four different preventive measures that may affect the surgical smoke exposure during total mastectomy surgery in the operating room of the General Surgery Department of a University HospitaL. The surgical resident, anaesthesiologist, anaesthesia technician and support staff included in the study did not consist of the same people due to the change in the work schedules. Blood and urine samples were collected from a team of seven people before and after surgery [7 volunteers × 2 (blood and urine before and after surgery) = 14 (14 blood analysis + 14 urine analysis) 14 × 5 surgery = 70 (70 blood analysis + 70 urine analysis)].
  Interventions: Other: surgical smoke affects

INTERVENTIONS:
Other: surgical smoke affects — The study, experimental type, was conducted to investigate the effects of five different methods on surgical smoke protection.
  Other Names: blood and urine samples

SUMMARY:
Background: Electrosurgery is used in almost all surgeries. The entire surgical team working in these operating rooms is exposed to surgical smoke. In the literature, there is no study examining the direct effect of surgical smoke on operating room staff and involving the entire surgical team in sampling.

Materials and Methods: This experimental-type study was conducted in the operating room of the Department of General Surgery of a University Hospital. In the study, the surgeries were completed with standard practice and four different protective measures that could affect surgical smoke exposure. Blood and urine samples were collected from the surgical team before and after the surgery. Consequently, 70 blood and 70 urine samples were collected. The Wilcoxon signed-rank test was used to compare pre- and post-operative analyses.

DETAILED DESCRIPTION:
2. MATERIALS AND METHODS 2.1 Design of the Study This was an experimental study. 2.2 Population and Sample of the Study Pre- and post-operative blood and urine samples of the surgical team (surgeon, surgical resident, anaesthesiologist, scrub nurse, circulating nurse, support staff and researcher), who worked in the standard practice, and the use of four different preventive measures that may affect the surgical smoke exposure during total mastectomy surgery in the operating room of the General Surgery Department of a University Hospital between January 2019 and December 2019 created the sample of the study. During the study process, the surgeon, scrub nurse, circulating nurse and researcher were ensured to be the same people in each surgery. The surgical resident, anaesthesiologist, anaesthesia technician and support staff included in the study did not consist of the same people due to the change in the work schedules. Blood and urine samples were collected from a team of seven people before and after surgery [7 volunteers × 2 (blood and urine before and after surgery) = 14 (14 blood analysis + 14 urine analysis) 14 × 5 surgery = 70 (70 blood analysis + 70 urine analysis)].

2.3 Collection of Study Data 2.3.1 Data Collection Tools The Surgery Data Collection Form, which was created by the researchers in line with the relevant literature (Romano et al. 2016, 2017, Ragde et al. 2014; Tseng et al. 2014, Lin et al. 2010, Hollmann et al. 2004) to evaluate the information about the surgery, was used to collect the data. Other data collection tools were the N95 and safety equipment, the RapidVac™ Smoke Evacuator system for smoke evacuation, as well as the pencil type (smoke extractor) and smoke tubing evacuators.

2.3.2 Data Collection Method Blood and urine samples of the surgical team were collected before the total mastectomy in five different situations listed below that may affect surgical smoke exposure.

After the surgery is completed with routine applications (without taking any measures for smoke evacuation), After completing the surgery with the use of special safety equipment (N95 mask, safety glasses and without any measures for smoke evacuation), After the evacuation of the smoke caused by the surgery with a wall-mounted aspirator, After the evacuation of the smoke caused by the surgery with a smoke tubing and After the evacuation of the smoke caused by the surgery with a smoke evacuation pencil.

The blood samples were kept in a transport bag that maintained the temperature range between 2 and 4 °C until they reached the laboratory and kept at -20 °C for analysis. Blood samples were evaluated in the laboratory for benzene, toluene, xylene and styrene.

Similarly, the urine samples were kept in a transport bag that maintained the temperature range between 2 and 4 °C until they reached the laboratory and kept at -20 °C for analysis. The urine samples were evaluated in terms of urinary metabolites benzene-phenol-TT muconic acid, toluene-hippuric acid-O, cresol, xylene-hippuric acid and phenol-phenol in the laboratory.

Blood and urine analysis in the study was performed by the Central Research Test and Analysis Laboratory Application and Research Center of the university of this study.

2.3.3 Evaluation and Analysis of Data The study data was evaluated using the IBM SPSS Statistics 25.0 Statistics program. The Wilcoxon signed-rank test was used to compare pre- and post-operative analyses. Moreover, 0.05 was accepted as significant.

Gas chromatography/mass spectrometry was used for the analysis of blood and urine samples of the surgical team.

2.4 Ethical Aspect of Study Permission (11.01.2018-E.11195) was obtained from the Clinical Research Ethics Committee of the university of this study. Also, written permission (29.01.2018-E27595) from the institution where the research was conducted as well as informed written consent from the participants in the study were obtained.

ELIGIBILITY:
Inclusion Criteria:

* Working in the operating room and smoke exposure during total mastectomy surgery
* Agree to participate in the study,

Exclusion Criteria:

* Working in the other operations
* Not wanting to give blood or urine sample

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-09-03 (Actual)

PRIMARY OUTCOMES:
Investigation of the preoperative and postoperative blood samples on Surgical Smoke Protection-Experimental Study | "an average of 6 month"
  Electrosurgery is used in almost all surgeries. The entire surgical team working in these operating rooms is exposed to surgical smoke. In the literature, there is no study examining the direct effect of surgical smoke on operating room staff and involving the entire surgical team in sampling. Blood and urine samples were collected from surgical team before and after surgery. Blood samples were evaluated in the laboratory for volatile organic compound (benzene, toluene, xylene and styrene etc.)
Investigation of the preoperative and postoperative urine samples on Surgical Smoke Protection-Experimental Study | "an average of 6 month"
  Electrosurgery is used in almost all surgeries. The entire surgical team working in these operating rooms is exposed to surgical smoke. In the literature, there is no study examining the direct effect of surgical smoke on operating room staff and involving the entire surgical team in sampling. Blood and urine samples were collected from surgical team before and after surgery. The urine samples were evaluated volatile organic compound (in terms of urinary metabolites benzene-phenol-TT muconic acid, toluene-hippuric acid-O, cresol, xylene-hippuric acid and phenol-phenol etc.) in the laboratory.

CONTACTS AND LOCATIONS:
Overall Officials: Burcak Sahin Koze, Mscn, Principal Investigator — Ege University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)